CLINICAL TRIAL: NCT05404633
Title: Usefulness and Acceptability of a Connected Ergocycle for the Elderly in a Clinical Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MP-31-2021-4146
Record Dates: First submitted 2021-07-08; First posted 2022-06-03 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradialytic exercise (patients) (Experimental): Participants in this group will use the tested device to perform a 30-minute session of aerobic training (cycling during hemodialysis) at 3-4/10 on the Borg scale of perceived exertion.
  Interventions: Device: Ergogycle prototype testing for acceptability
- Acute care exercise (patients) (Experimental): Participants in this group will use the tested device to perform 2 x 10-minute of aerobic training (cycling in the hospital) interspersed with a 5-minute break. Exercise intensity will be of 2/10 on the Borg scale of perceived exertion (around 3 +/- 2 watts at 20 rpm).
  Interventions: Device: Ergogycle prototype testing for acceptability

INTERVENTIONS:
Device: Ergogycle prototype testing for acceptability — The objective was to assess the acceptability of the ergogycle prototype (device) while used in a clinical settings by both the patients and the professionals.

SUMMARY:
Hospitalizations are harmful to patients. Without a proper intervention, it will lead to a permanent decline in physical function, especially among frail individuals. Ultimately, this will worsen quality of life, as well as the cognitive and functional status of affected elderly people, which will arguably reduce functional independence, increase post-discharge institutionalization and death among frail older adults. It is known that patients receiving early physical evaluation and rehabilitation (in the 24 hours following admission) improves post-discharge orientation, decreases delirium and the need of acute care. The rehabilitation often involves ergocycles, but commercially available devices are expensive and often hard to move, to set up in hospital bed and lack connectivity.

In this context, a connected ergocycle prototype which has a number of desired characteristics, including low production cost, relatively light and easy to move and with internet connectivity. The goal of this study is thereby to assess the usefulness and acceptability of the prototype with health professionals involved in physical rehabilitation and patients receiving said rehabilitation.

ELIGIBILITY:
Inclusion Criteria :

* > 55 years old
* receiving treatments for terminal renal insufficiency at least 3 times a week, for at least 3 months (hemodialysis; HD) or under mechanical ventilation for less than 72 hours, and that should last for at least 24 more hours (intensive unit care; ICU)
* Physically independent outside HD or before admission (ICU) (≥ 70 on the Barthel index)
* with medical clearance (HD : nephrologist; ICU : intensivist)

Exclusion Criteria:

* unable to walk without assistance (before ICU admission)
* diagnosed neurocognitive decline
* recent hemiarthroplasty for a hip fracture that causes a limitation in the flexion of the hip during pedaling
* already involved in another study

Exclusion Criteria Specific for ICU Patients :

* neuromuscular disorder affecting the weaning from mechanical ventilator support
* pathologic fracture or unstable cervical spine fracture
* hospitalized for more than 7 days
* COVID-19 positive
* reported as moribund by the intensivist

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the device | up to 1 hour after the exercise session for both the patients and professionals
  Questionnaire based on the unified theory of acceptance and use of technology

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec, Canada